CLINICAL TRIAL: NCT00572351
Title: The Effects of Red Wine and White Wine on Blood Estrogen and Progesterone Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director of the Barbra Streisand Women's Heart Center at Cedars-Sinai Medical Center, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB 6110
Record Dates: First submitted 2007-01-11; First posted 2007-12-13 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Wine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red Wine (Active Comparator)
  Interventions: Other: Red Wine
- White Wine (Active Comparator)
  Interventions: Other: White Wine

INTERVENTIONS:
Other: Red Wine — 8 ounces of assigned beverage (red wine) each evening and abstinence from any other alcoholic beverages, grape juice, grapes, or raisins.
  Arms: Red Wine
Other: White Wine — 8 ounces of assigned beverage (white wine) each evening and abstinence from any other alcoholic beverages, grape juice, grapes, or raisins.
  Arms: White Wine

SUMMARY:
Healthy pre-menopausal women will be recruited in order to test the effects of red wine and white wine on blood estrogen and progesterone levels. The women will be randomized and rotated through two different treatments (red wine, white wine). Estrone and estradiol are hormones in the category of estrogens. It is known that the bodies of both men and women may convert (or aromatize) a certain amount of naturally occurring testosterone into estrogen. Aromatase inhibitors have been used to prevent this conversion, or aromatization, of testosterone into estrogen, in the treatment of estrogen-dependent breast cancer in women. This inhibition leads to a marked decrease in estrogen (estradiol and estrone) levels. Naturally occurring aromatase inhibitors include grapes, grape juice, and red, but not white wine. The aromatase inhibitory effects are attributed to wine phytochemicals and not to alcohol. Based upon this information, the investigators will monitor the estrogen levels at various phases in the menstrual cycles of women since hormone levels naturally vary throughout the menstrual cycle. Several epidemiologic studies have found that there is a correlation with moderate to high levels of alcohol consumption and breast cancer. Therefore, study participants will be asked to drink only a eight ounces of wine which should have minimal or no risk for the development of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. female
2. pre-menopausal with regular ovulatory cycles for 12 months prior to the study
3. willingness and ability to participate in study requiring alcohol consumption
4. in general good health
5. BMI of 18.5-35
6. on regular, unrestricted diet
7. not currently, or within the past 3 months, using oral contraceptives or other hormone replacement therapy

Exclusion Criteria:

1. male
2. irregular menstrual cycles or vasomotor symptoms within the last 12 months
3. pregnant (or breast feeding)
4. any hormone therapy including phytoestrogens, oral contraceptives, SERMs (selective estrogen receptor modulators), or androgens (or precursors) for three months prior to the study
5. history of alcohol abuse
6. history of any estrogen-dependent neoplasia
7. high intake of dietary soy products
8. Minors < age 21 years

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
blood estrogen and progesterone levels | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Glenn D Braunstein, MD, Principal Investigator — Cedars Sinai Medical Cneter
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shufelt C, Merz CN, Yang Y, Kirschner J, Polk D, Stanczyk F, Paul-Labrador M, Braunstein GD. Red versus white wine as a nutritional aromatase inhibitor in premenopausal women: a pilot study. J Womens Health (Larchmt). 2012 Mar;21(3):281-4. doi: 10.1089/jwh.2011.3001. Epub 2011 Dec 7. PMID 22150098